CLINICAL TRIAL: NCT03442387
Title: Framing of Numerical Information in Cochrane Summaries: a Randomized Controlled Trial
Brief Title: Framing of Numerical Information in Cochrane Summaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Ivan Buljan, Research Assistant, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Grant No. IP-2014-09-7672
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Health Literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive frame (Experimental): The numerical expressions were presented in a positive way: e.g. treatment was successful for 4 out of 10 persons.
  Interventions: Other: Frame of numerical information
- Negative frame (Experimental): The numerical expressions were presented in a negative way: e.g. treatment was unsuccessful for 6 out of 10 persons.
  Interventions: Other: Frame of numerical information

INTERVENTIONS:
Other: Frame of numerical information — Each group received only one frame of information.

SUMMARY:
The aim of the study was to conduct three different parallel randomized controlled trials to assess how the different framing of Cochrane summary information (positive vs negative framing of health information) affects affect the perception of the efficacy and intention for use of the described treatment.

DETAILED DESCRIPTION:
The aim of the study was to conduct three different parallel randomized controlled trials to assess how the different framing of Cochrane summary information (positive vs negative framing of health information) affects affect the perception of the efficacy and intention for use of the described treatment.

ELIGIBILITY:
Inclusion Criteria:

* First year medical students

Exclusion Criteria:

* Those who have failed first year and have to repeat it.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Perception of effectiveness | Immediately after reading
  One item on Likert type scale from 1-10, higher score indicates the higher perceived effectiveness.

SECONDARY OUTCOMES:
Desire to use the described treatment | Immediately after reading
  One item on Likert type scale from 1-10, higher score indicates the greater desire to use the described treatment.
Desire that treatment is prescribed by family doctor | Immediately after reading
  One item on Likert type scale from 1-10. Higher score indicates the greater desire that treatment is prescribed by family doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Buljan, MPsy, Principal Investigator — University of Split, School of Medicine
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Available upon request from principal investigator.
Supporting Information: SAP

REFERENCES:
- [Derived] Buljan I, Tokalic R, Roguljic M, Zakarija-Grkovic I, Vrdoljak D, Milic P, Puljak L, Marusic A. Framing the numerical findings of Cochrane plain language summaries: two randomized controlled trials. BMC Med Res Methodol. 2020 May 6;20(1):101. doi: 10.1186/s12874-020-00990-4. PMID 32375659